CLINICAL TRIAL: NCT01072643
Title: The Pharmacodynamics, Safety, and Pharmacokinetics of Sedation With Dexmedetomidine in Children Undergoing Hemodynamic Cardiac Catheterization With Special Reference to the Pulmonary Vascular Bed
Brief Title: Sedation With Dexmedetomidine During Cardiac Catheterization
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Study was terminated due to increased PVR in one subject from T0-T1 reaching the level of a predetermined stopping rule
Sponsor: Aruna Nathan (Other)
Collaborators: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor-Investigator, Aruna Nathan, Attending Physician, Children's Hospital of Philadelphia
Organization: Children's Hospital of Philadelphia (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-007076
Record Dates: First submitted 2010-02-15; First posted 2010-02-22 (Estimated); Results first posted 2014-09-08 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Pulmonary Hypertension
Keywords: Sedation; Pulmonary Hypertension; Pediatric; Cardiac Catheterization; Pulmonary Vascular Resistance
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dexmedetomidine (Experimental): To study safety of DEX with regard to effect on PVR; There will be 3 study groups (n=8 per group). The groups will be based on DEX doses as follows- Group 1 - Bolus 1 mcg/kg followed by infusion 0.7 mcg/kg/hr Group 2 - Bolus 1.5 mcg/kg followed by infusion 1.05 mcg/kg/hr Group 3 - Bolus 2 mcg/kg followed by infusion 1.4 mcg/kg/hr
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — This is a single center, dose escalation study of Dexmedetomidine in pediatric subjects with pulmonary hypertension (PVR>4WU) undergoing hemodynamic cardiac catheterization and vasoreactivity drug testing. Cohorts of 8 evaluable subjects will receive dose level 1, dose level 2, or dose level 3 of Dexmedetomidine.
  Other Names: Precedex

SUMMARY:
Clinical dose escalation drug trial to evaluate the effect of 3 different doses of dexmedetomidine on the pulmonary vascular bed in pediatric subjects with elevated pulmonary vascular resistance (PVR). The study will be conducted in 2 parts, with part 1 incorporating stopping rules to optimize safety of the drug in this population. The second part of this study will evaluate if the lowest safest dose, as determined in part 1, is adequate to provide effective sedation during a cardiac catheterization procedure.

DETAILED DESCRIPTION:
Clinical dose escalation drug trial to evaluate the effect of 3 different doses of dexmedetomidine on the pulmonary vascular bed in pediatric subjects with elevated pulmonary vascular resistance. The study will be conducted in 2 parts, with a pilot phase incorporating stopping rules to optimize safety of the drug in this population. Study subjects will include pediatric subjects with Pulmonary Hypertension (PHTN).

Part 1: This will be the dose escalation phase of the study. Twenty four evaluable subjects will be enrolled. Subjects will include pediatric subjects with pulmonary hypertension (PVR>4WU) undergoing hemodynamic cardiac catheterization and vasoreactivity drug testing. Cohorts of 8 evaluable subjects will receive dose level 1, dose level 2, or dose level 3 of Dexmedetomidine (DEX). The dose will be escalated to the next dose of DEX once all subjects have been enrolled in the preceding DEX dose cohort, and safety has been established at that level. Inadequate sedation despite the highest dose of DEX at each level will be considered a treatment failure on an intention to treat basis. Part 2: This part of the study will be conducted after the pilot phase is safely completed, and the full complement of subjects will be recruited.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with a diagnosis of pulmonary hypertension
2. Procedure - Planned cardiac catheterization procedure with spontaneous ventilation and natural airway
3. Patients who want sedation or general anesthetic for the procedure.
4. Age: Subjects ≥8 years and < 21 years
5. Adequate Renal Function defined As:Serum creatinine ≤ 1 mg/dL
6. Adequate Liver Function defined As:Total bilirubin ≤ 1.5 mg/dL alanine aminotransferase (ALT) ≤ 2 times the upper limit of normal
7. Informed Consent: All parents or legal guardians must sign a written informed consent.
8. Signed assent when developmentally appropriate
9. Negative pregnancy test in menstruating females and all females ≥ 12 yr

Exclusion Criteria:

1. Refusal of Informed Consent/Assent
2. Subjects with single ventricle physiology
3. Pregnant or lactating females
4. Subjects with syndromes e.g. Trisomy 21 will be excluded due to variability in pharmacodynamic responses and airway instability during sedation
5. Inappropriate clinical or developmental status to undergo cardiac catheterization under conditions of spontaneous ventilation with a natural airway
6. Second or third degree heart block
7. Moderate - severe right ventricular dysfunction/failure
8. Subjects who, in the opinion of the investigator, are not appropriate candidates for an investigational drug study e.g. behavioral or anxiety disorders, inability to lie supine
9. Concomitant Medications - Investigational Drugs: Subjects who have received another investigational drug protocol 30 days prior to enrollment in this study
10. Subjects who in the opinion of the investigator may be non compliant with study schedules or procedures.
11. Non-English speaking subjects will be excluded due to need for direct communication from clinical and study staff during study procedures and the ability to complete study tools.

Ages: 8 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4 (Actual)
Dates: Start 2010-03; Primary Completion 2013-03 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aruna T Nathan, MBBS, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 22 patients were screened, but 18 were determined to be not feasible, only 4 participants were enrolled and started the study at drug level 1 (bolus of 1mcg/kg and infusion at 0.7mcg/kg/hr); There was no escalation to either dose level 2 or dose level 3 as we did not reach enrollment target of 8 subjects in dose level 1
Groups:
- Dexmedetomidine (DEX) 1 mcg/kg Bolus: To study safety of Dexmedetomidine (DEX) with regard to effect on PVR; There will be 3 study groups (n=8 per group). The groups will be based on DEX doses as follows- Group 1 - Bolus 1 mcg/kg followed by infusion 0.7 mcg/kg/hr Group 2 - Bolus 1.5 mcg/kg followed by infusion 1.05 mcg/kg/hr Group 3 - Bolus 2 mcg/kg followed by infusion 1.4 mcg/kg/hr
  Dexmedetomidine: This is a single center, dose escalation study of Dexmedetomidine in pediatric subjects with pulmonary hypertension (PVR>4WU) undergoing hemodynamic cardiac catheterization and vasoreactivity drug testing. Cohorts of 8 evaluable subjects will receive dose level 1, dose level 2, or dose level 3 of Dexmedetomidine.
Period: Overall Study
Arm/Group | Dexmedetomidine (DEX) 1 mcg/kg Bolus
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Children with PHTN who received Dex sedation for cardiac catheterization.
Arm/Group | Dexmedetomidine
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 1

OUTCOME MEASURES:

1. Primary Outcome: The Primary Endpoint Will be the Change in PVR in Wood Units
Description: Pulmonary vascular resistance (PVR) in Wood units calculated during cardiac catheterization;
Time Frame: For each subject PVR will be measured by cardiac catheterization at T0 ( baseline measurement) , after DEX bolus (T1) which is given over 10 minutes and after 30 mins after start of the DEX infusion (T2) - Maximum upto 4 hours
Measure: Number; unit: wood units
Groups:
- Subject 1; Subject 2; Subject 3; Subject 4: Pulmonary vascular resistance (PVR) in Wood units calculated during cardiac catheterization
Arm/Group | Subject 1 | Subject 2 | Subject 3 | Subject 4
Number analyzed (Participants) | 1 | 1 | 1 | 1
wood units
  T0 | 8.9 | 13.7 | 5.45 | 8.57
  T1 | 9.7 | 15.5 | 6.52 | 13.18
  T2 | 7.1 | 15.5 | 7.0 | 2.27

2. Secondary Outcome: Efficacy of Sedation With DEX
Description: The study was terminated early due to increased pulmonary vascular resistance (PVR) in one subject from To-T1 reaching the level of a predetermined stopping rule. Investigators suggested that it is premature to conclude that DEX does not adversely affect PVR
Time Frame: Subjects will participate in a dose escalation study which will define minimal effective dose that results in effective sedation in ≥ 7 out of 8 patients in that dose cohort. Maximum upto 4 hours
Population: The study was terminated early due to increased pulmonary vascular resistance (PVR) in one subject from To-T1 reaching the level of a predetermined stopping rule. Investigators suggested that it is premature to conclude that DEX does not adversely affect PVR.
Groups:
- Subject 1; Subject 2; Subject 3; Subject 4: Efficacy of sedation with DEX
Arm/Group | Subject 1 | Subject 2 | Subject 3 | Subject 4
Number analyzed (Participants) | 0 | 0 | 0 | 0

3. Secondary Outcome: Quantify the Effect of DEX on PVR in Pediatric Subjects With Pulmonary Hypertension (PHTN) and Its Dependence on Baseline PVR
Description: as for outcome 2
Time Frame: Every individual patient will be studied over maximum of 4 hours during the dose escalation phase. This part of the study will be completed in 1 year
Population: as for outcome 2
Groups:
- Subject 1; Subject 2; Subject 3; Subject 4: Quantify the effect of DEX on PVR in pediatric subjects with pulmonary hypertension and its dependence on baseline PVR
Arm/Group | Subject 1 | Subject 2 | Subject 3 | Subject 4
Number analyzed (Participants) | 0 | 0 | 0 | 0

4. Secondary Outcome: Obtain Pharmacokinetic Data in This Population
Description: as for outcome 2
Time Frame: 6 hours
Population: as for outcome 2
Groups:
- Subject 1; Subject 2; Subject 3; Subject 4: Obtain pharmacokinetic data in this population
Arm/Group | Subject 1 | Subject 2 | Subject 3 | Subject 4
Number analyzed (Participants) | 0 | 0 | 0 | 0

5. Secondary Outcome: Demonstrate That DEX is a Safe Sedative in Pediatric Subjects With PHTN
Description: as for outcome 2
Time Frame: 24 hours
Population: as for outcome 2
Groups:
- Subject 1; Subject 2; Subject 3; Subject 4: Demonstrate that DEX is a safe sedative in pediatric subjects with PHTN
Arm/Group | Subject 1 | Subject 2 | Subject 3 | Subject 4
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Dexmedetomidine
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes